CLINICAL TRIAL: NCT06289244
Title: Correlation Between Muscle Strength and Thickness in Critically Ill Patients: an Observational Prospective Study
Brief Title: Correlation Between Muscle Strength and Thickness in Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Veronica Rossi, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 6597
Record Dates: First submitted 2024-02-04; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness; Muscle Weakness
Keywords: Intensive Care Units; Respiration, Artificial; Limb Muscle Assessment; Diaphragm thickness; Respiratory Distress Syndrome
MeSH Terms: conditions — Critical Illness; Muscle Weakness; Respiratory Aspiration; Respiratory Distress Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — The thickness of the diaphragm and quadriceps will be assessed using bedside ultrasound, utilizing a 13-6 MHz cm linear probe. The measurement of the right hemidiaphragm's end-expiratory thickness will be conducted via diaphragm ultrasound. For accurate positioning, the ultrasound probe will be placed along the right anterior axillary line, specifically between the ninth and tenth intercostal spaces, in a sagittal oblique orientation. To enhance measurement consistency, the probe's position on the skin will be marked.
  To ascertain accuracy, the operator will conduct each measurement three times, and the mean of these three values will be used for analysis. Similarly, for diaphragmatic assessment and peripheral assessments (Qthick and CSA) of the lower limbs, the examination areas will be demarcated on the skin with a dermatographic pen, ensuring measurement reproducibility over different timepoints.
Diagnostic Test: Muscle strength measurement — The assessment of limb muscle strength in this study will be conducted using the Medical Research Council (MRC) Score. For a more precise evaluation of quadriceps strength, a dynamometer will be employed.
  Furthermore, the study will incorporate an invasive method for gauging inspiratory muscle strength, utilizing the negative inspiratory force (NIF) metric. Post-extubation, the maximum inspiratory pressure (MIP) will be determined using an electronic manometer. Three separate MIP measurements will be executed, and the highest reading among these will be recorded as the definitive measurement.

SUMMARY:
Mechanical ventilation (MV) is associated with adverse outcomes in ventilated patients, and impact of MV-induced diaphragm changes are still unclear.

The objective of this prospective observational study is to assess muscle thickness and strength, specifically in limb muscles such as the quadriceps, among critically ill patients who undergo extended mechanical ventilation during their Intensive Care Unit (ICU) stay.

The primary inquiries this study seeks to address are:

* Is there an association between muscle thickness and strength in the limbs of critically ill patients undergoing prolonged MV?
* How much thickness and strength variation can be expected in respiratory and limb muscles in critically ill patients undergoing prolonged MV?

DETAILED DESCRIPTION:
The methodology for measuring the thickness of the diaphragm and quadriceps involves the use of bedside ultrasound. In terms of diaphragmatic assessment, to ensure consistency over multiple timepoints, the areas of the lower limbs evaluated (Quadriceps thickness, Qthick and Cross section area, CSA) will be marked on the skin using a dermatographic pen during the peripheral assessments.

Muscle strength in the limbs will be assessed utilizing the Medical Research Council (MRC) Score, specifically in patients who are awake and cooperative (RASS 0 +/- 1). Additionally, a dynamometer will be employed for the precise measurement of quadriceps strength, serving as the gold standard.

The timeline for data collection during the observational period is structured as follows:

T1: 48-72 hours from the start of invasive MV after intubation T2: At the initial trial in pressure support mode. T3: Immediately prior to extubation. T4: Before discharge from the Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Intubated patients on mechanical ventilation presumably for 48 hours;
* Informed consent

Exclusion Criteria:

* Contraindication (absolute or relative) to assessment: acute bleeding, multiple fractures or trauma, spinal instability;
* Hemodynamic instability during assessment;
* ICU admission due to thoracic surgery, including lung transplant patients;
* History of preexisting neuromuscular diseases;
* History of preexisting functional impairment;
* Pheripheral Neural disease;
* Cervical spine injury;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Intensive Care Unit (ICU) who are expected to need mechanical ventilation for at least 48 hours following ARDS.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between quadriceps strength and thickness | The assessment will be perform at 48-72 hours from start of invasive MV after intubation, at the initial trail in pressure support mode, at immediately prior to extubation and at discharge from the Intensive Care Unit (assessed up to 5 months)
  Degree of correlation between quadriceps strength, measured via handheld dynamometer (strength in Newton), and thickness, measured using ultrasound (thickness in cm).

SECONDARY OUTCOMES:
Quadriceps strength | The assessment will be perform at 48-72 hours from start of invasive MV after intubation, at the initial trail in pressure support mode, at immediately prior to extubation and at discharge from the Intensive Care Unit (assessed up to 5 months)
  Mean difference of quadriceps strength along ICU stay period
Quadriceps thickness | The assessment will be perform at 48-72 hours from start of invasive MV after intubation, at the initial trail in pressure support mode, at immediately prior to extubation and at discharge from the Intensive Care Unit (assessed up to 5 months)
  Mean difference of quadriceps thickness along ICU stay period
Diaphragm thickness | The assessment will be perform at 48-72 hours from start of invasive MV after intubation, at the initial trail in pressure support mode, at immediately prior to extubation and at discharge from the Intensive Care Unit (assessed up to 5 months)
  Mean difference of diaphragm thickness along ICU stay period
Diaphragm strength | The assessment will be perform at 48-72 hours from start of invasive MV after intubation, at the initial trail in pressure support mode, at immediately prior to extubation and at discharge from the Intensive Care Unit (assessed up to 5 months)
  Mean difference of diaphragm thickness along ICU stay period
Time to reach the sitting position | The assessment will be perform at 48-72 hours from start of invasive MV after intubation, at the initial trail in pressure support mode, at immediately prior to extubation and at discharge from the Intensive Care Unit (assessed up to 5 months)
  Mean difference of number of days required to reach the sitting position

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Rossi, MSc, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Umbrello M, Guglielmetti L, Formenti P, Antonucci E, Cereghini S, Filardo C, Montanari G, Muttini S. Qualitative and quantitative muscle ultrasound changes in patients with COVID-19-related ARDS. Nutrition. 2021 Nov-Dec;91-92:111449. doi: 10.1016/j.nut.2021.111449. Epub 2021 Aug 15. PMID 34583135
- [Background] Dres M, Dube BP, Mayaux J, Delemazure J, Reuter D, Brochard L, Similowski T, Demoule A. Coexistence and Impact of Limb Muscle and Diaphragm Weakness at Time of Liberation from Mechanical Ventilation in Medical Intensive Care Unit Patients. Am J Respir Crit Care Med. 2017 Jan 1;195(1):57-66. doi: 10.1164/rccm.201602-0367OC. PMID 27310484